CLINICAL TRIAL: NCT03912311
Title: Comparison Between Diagnostic Performances of Auscultation and Ultrasonography Respect of Fiberoptic Bronchoscopy in the Valuation of Positioning of Endotracheal Double-lumen Tube in Elective Thoracic Surgery
Brief Title: Auscultation, Lus, Fob In Olv (ALFIO)
Acronym: ALFIO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Elena Giovanna Bignami, Professor of Anesthesiology, University of Parma
Other Study IDs: ALFIO2019
Record Dates: First submitted 2019-04-05; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Thoracic Anesthesia; Lung Ultrasound; Left Double-lumen Tube; Selective Bronchial Intubation; One-lung Ventilation; Auscultation; Flexible Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will be to demonstrate that, in patients undergoing elective thoracic surgery, lung ultrasound (LUS) in OR is more sensitive, specific and accurate method than thoracic auscultation, for the evaluation of OLV. The aim of the study is to demonstrate how lung ultrasound can be considered an attractive alternative to the routine use of fiberbronchoscope as a first line diagnostic tool to verify the correct position of left double lumen tube.

DETAILED DESCRIPTION:
Most procedures in thoracic surgery require exclusion from ventilation of the lung undergoing surgery. One-lung ventilation (OLV), it is obtained mainly through the placement of a bi-lumen tube (DLT) in the patient's airway. A frequent complication that occurs during OLV it's unrecognized bad positioning of the DLT which can lead to serious complications such as hypoventilation, hypoxemia, not optimal collapse of the operated lung and damage to the trachea or main bronchi.

The latest SIAARTI recommendations (2009) advocate in all patients use of fiberbronchoscope (FOB) to control and correct the positioning of the DLT (gold standard) after the orotracheal intubation and after the positioning in lateral decubitus. The usual clinical practice expects to performing lung exclusion tests by auscultation of the 2 hemithorax in succession. But the scientific evidence shows how this practice has a poor sensitivity and specificity in assessing the correct positioning of the left DLT (LDLT). From literature, as from everyday clinical experience, it is known that FBS cannot always be performed Finally, the research wants to shed light how the fiberoptic bronchoscopy (FBS) is an invasive maneuver that is not free from serious complications (mucosal lesions and infections).

Ultrasound (US) over the last 15 years has made an important contribution to the assessment and management of the airways. US quickly and effectively are able to show the excursion of the diaphragm and pleura, qualitative and quantitative indicators of lung expansion. If the endotracheal tube is in the correct position, a bilateral and symmetrical movement of the domes of each hemi-diaphragm (B-Mode and M-mode) can be appreciated, while in the intercostal window, the so-called "lung-sliding" will be visible. In the absence of ventilation, the diaphragmatic excursion and the "lung-sliding" will not be detectable in the explored hemi-thorax.

Although FBS remains the gold standard for controlling the correct position of LDLT under thoracic anesthesia, and is often crucial as a guide to its repositioning, from the researchers point of view, the use of FOB may not be routinely necessary in all patients, but its use could be reserved for selected cases in which the positioning itself is difficult or in case of intraoperative displacement. Primary objective is to demonstrate how, in patients undergoing elective thoracic surgery, lung ultrasound (LUS) to the operating room is a more sensitive, specific and accurate method than thoracic auscultation, for the evaluation of OLV. LUS is a non-invasive, safe and free from side effects technique that can be performed at the patient's bed. The study aims to demonstrate how LUS can be considered an attractive alternative to the routine use of FOB as a first line diagnostic tool to verify the correct position of LDLT.

For each surgical procedure 3 researchers will participate, each with a specific independent role: the auscultation researcher (AR), which will have the task of performing the oral-tracheal intubation and auscultation with phonendoscope pre-and post-induction of general anesthesia and after positioning the patient in lateral decubitus; the ultrasound researcher (UR), i.e. the anesthesiologist who will perform the pre- and post-induction of the AG ultrasound evaluation and after positioning the patient in lateral decubitus; the Fiberscope Researcher (FR), whom will perform the fibrobroncoscopic verification of the LDLT at the end of the clinical and ultrasound assessment and after the positioning in lateral position. He will reposition the endotracheal tube in case of mal positioning or intra-operative displacement of the same.

Upon the arrival of the patients in the operating room, and after applying the standard operative monitoring for the planned surgery, the AR will perform a preliminary thoracic auscultation, in order to verify the presence of normal lung sounds in spontaneous breathing. The UR will perform a preliminary thoracic ultrasound scanning, in order to verify the presence of long sliding (LS) and diaphragmatic displacement (DD). Then, after the positioning of adequate venous accesses and eventually a medium-thoracic peridural catheter, AR will proceed to induce general anesthesia. Patients will undergo video-thoracoscopy or thoracotomy operations that require mono-pulmonary ventilation (OLV) for each part or for the entire duration of the operation. The choice of the appropriate LDLT size will be made on the basis of Brodsky's anthropometric criteria. After sedation and curarization, direct laryngoscopy will be performed with a Macintosh blade and patients will be intubated with a left bi-lumen (LDLT) Carlens or Robertshaw tube by the AR, after that he will also perform auscultation. After inflating the tracheal cuff and verifying the symmetricity of the vesicular murmure on both pulmonary fields in two pre-established points per side (apex = II-III intercostal space on the hemiclavicular; base = V intercostal space on the middle axilla), the bronchial cuff will be inflated and the auscultation repeated by first clamping the tracheal lumen and then the bronchial lumen. If the LDLT is correctly positioned the MV will be present at the apex and base of the ventilated lung and absent in the contralateral points of the excluded lung. Otherwise the LDLT will be considered wrongly positioned and the AR will have 3 attempts to reposition the device. The AR will record the results of the verification carried out on the CRF and will leave its role in the OR at the UR. The latter, using a 6-13 MHz linear ultrasound probe, will evaluate, in B-mode and M-mode, the presence / absence of the LS and the LP at the level of the II-III intercostal space on the hemiclavicular, while with a convex ultrasound probe 3,5-5 MHz placed orthogonally to the costal arch on the anterior axillary line, the diaphragmatic displacement will be searched and measured. The bi-lumen tube will be considered correctly positioned in the presence of LS and DD in the ventilated lung and in their absence in the excluded lung. Otherwise the LDLT will be considered wrongly positioned.

The UR will record the results of the verification carried out on the CRF and will leave its position in the operating room at the FR. Finally, the correct positioning of the LDLT will be verified with FOB from the FR and eventually repositioned. The bronchoscope will be introduced into the tracheal lumen and get throw until it reaches just beyond the tracheal hole. The correct vision foresees: the carena on the sagittal plane and on the right the orifice of the right main bronchus, while on the left, the dome of the bronchial cap occupying the orifice of the left main bronchus. The final judgment of the FR will be: "correct positioning", "malposition", "critical malposition". Each researcher will not know the outcome of the verification carried out by the other 2 researchers.

Once the correct positioning of the LDLT has been verified, if necessary by the surgical requirements, the patient will be placed in lateral position and a new pulmonary exclusion test will be performed. AR, UR and FR will perform again the lung test exclusion, reporting in the CFR the results of the new evaluations. These assessments will be made by the same researchers who performed the previous assessments.

During the intra-operative phase the ventilation and maintenance of general anesthesia will be set according to the standard clinical practice and data will be reported in the appropriate section of the CFR concerning vital and ventilation parameters, the time required for pulmonary exclusion tests, any displacement of the LDLT and any surgical and non-surgical complications.

At the end of the surgical procedure, after optimization of the analgesia and according to the patient's needs, the patient will be extubated in the operating room or transfered in the the post-operative intensive care unit. The collection of clinical data will continue in the post-operative period until the hospital discharge of the patient enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age > 18 years
* Patients who underwent elective thoracic surgery (video-assisted thoracic surgery or open thoracotomy) requiring lung isolation and endotracheally intubation by LDLT

Exclusion Criteria:

* Not signed informed consent
* Age < 18 years
* Previous history of thoracic surgery
* Planned use of right double lumen tube
* Pleural diseases: pleural spill, pneumothorax, mesothelioma, previous pleurodesis
* Neuromuscular disease with proved diaphragmatic disfunction
* Thoracic subcutaneous emphysema
* Difficult endotracheally intubation or more than 3 attempts made by an experienced anesthesiologist or alternative device use
* Pregnancy
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent elective thoracic surgery (video-assisted thoracic surgery or open thoracotomy) requiring lung isolation and endotracheally intubation by left double lumen tube
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-04-02 (Estimated); Primary Completion 2020-04-02 (Estimated); Study Completion 2020-06-02 (Estimated)

PRIMARY OUTCOMES:
To compare trans- thoracic ultrasound method and auscultation in left selective intubation with LDLT, considering them as an alternative to fiberoptic bronchoscope use. | Through study completion, an average of 1 years
  Sensitivity, specificity and accuracy of ultrasound method and auscultation method as technique to verify LDLT correct placement, checked with fiberoptic bronchoscope.

SECONDARY OUTCOMES:
Incidence of LDLT malpositioning | Through study completion, an average of 1 years
Incidence of LDLT displacements after lateral positioning and during surgery | Through study completion, an average of 1 years
Incidence of intra- and post-operating complications | Through study completion, an average of 1 years
Presence/absence of lung sliding throw ultrasound scan in case of correct/incorrect position of LDLT | Through study completion, an average of 1 years
Presence/absence of lung pulse throw ultrasound scan in case of correct/incorrect position of LDLT | Through study completion, an average of 1 years
Measure of diaphragmatic displacement throw ultrasound scan in spontaneous breath and in mechanical ventilation | Through study completion, an average of 1 years
Evaluation time to perform lung ultrasound scansion during lung exclusion test | Through study completion, an average of 1 years
Evaluation time to perform auscultation during lung exclusion test. | Through study completion, an average of 1 years
Evaluation time to verifing of position of LDLT with FOB | Through study completion, an average of 1 years
Incidence of ICU admission (planned or unplanned) | Through study completion, an average of 1 years
ICU and Hospital length of stay | Through study completion, an average of 1 years
Incidence of mortality | Through study completion, an average of 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Michela Tosi, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Massimo Maffezzoni, MD, Principal Investigator — Università di Parma; Piercarlo Cottone, MD, Principal Investigator — Università di Parma; Stefania Lepori, MD, Principal Investigator — Università di Parma; Valentina Bellini, MD, Principal Investigator — Università di Parma
Locations (1):
- Azienda Ospedaliera-Universitaria di Parma, Parma, Italy